CLINICAL TRIAL: NCT06764251
Title: A Single-centre Phase II Clinical Study of Tislelizumab Combined with SOX Regimen in the Treatment of Locally Advanced Gastric Cancer/gastroesophageal Junction Adenocarcinoma
Brief Title: Tislelizumab Combined with SOX Regimen in the Treatment of Locally Advanced Gastric Cancer/gastroesophageal Junction Adenocarcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Liaoning Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Zheng Zhichao, Offices Director, Liaoning Cancer Hospital & Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NeoGC-01
Record Dates: First submitted 2024-12-17; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Gastric/Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tislelizumab + SOX (Experimental)
  Interventions: Drug: Tislelizumab + SOX

INTERVENTIONS:
Drug: Tislelizumab + SOX — tislelizumab combined with SOX

SUMMARY:
This study is to evaluate the efficacy of neoadjuvant long-term treatment with tislelizumab in combination with SOX in the treatment of locally advanced gastric/gastroesophageal junction adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to participate in this study, able to sign the informed consent form, and with compliance;
2. No gender restriction, aged ≥18 and ≤70 years (at the time of signing the informed consent form);
3. ECO score of 0-1;
4. Estimated survival ≥6 months;
5. HER-2 negative;
6. Central laboratory confirmed PD-L1 expression in the, with a combined positive score (CPS) ≥1;
7. Histological and radiological assessment confirmed as advanced gastric cancer (GC) or gastroesal junction (GEJ) adenocarcinoma, with a clinical stage of cT3-T4aN M0;
8. Pre-enrollment by the attending physician to determine eligibility for R0 resection with curative intent;
9. Good cardiac function. Patients with underlying ischemic, valvular disease, or other severe heart disease should have a preoperative assessment by a cardiologist if there are clinical indications;
10. No prior cytotoxic or targeted, no prior partial or complete esophagogastric tumor resection;
11. Negative for hepatitis B surface antigen (HBsAg) and hepatitis core antibody (HBcAb). If HBsAg is positive or HBcAb is positive, then the hepatitis B virus deoxyribonucleic acidHBV-DNA) must be <1000 copies/mL or <200 IU/mL or <the upper limit of normal (ULN) at research center to be eligible;
12. Negative for hepatitis C virus (HCV) antibody;
13. Normal major organ function, as defined by the criteria (within 14 days before the first dose, without transfusions, albumin, recombinant human thrombopoietin, or colony-stulating factor (CSF) treatment): Blood routine examination: Hemoglobin (Hb) ≥90g/L; absolute neutrophil count (ANC ≥1.5×109/L; platelets (PLT) ≥80×109/L; Biochemical examination: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN (≤5×ULN liver metastasis); total bilirubin (TBIL) ≤1.5×ULN (≤3×ULN for Gilbert's syndrome); seruminine (Cr) ≤1.5×ULN, or creatinine clearance rate ≥60mL/min; Coagulation function: Activated partialboplastin time (APTT), international normalized ratio (INR), and prothrombin time (PT) ≤1.5×ULN; Dpler ultrasound assessment: Left ventricular ejection fraction (LVEF) ≥50%; Normal thyroid function, defined as thyroid-stimulating hormone (T) within the normal range. If baseline TSH is out of range, patients with total T3 (or FT3) and FT4 within the normal range also be included; Clinical judgment by the doctor that organ function is sufficient.
14. Fertile subjects must use appropriate contraception during the study and for 20 days after the study ends, have a negative serum pregnancy test within 7 days before enrollment, and must not be breastfeeding

Exclusion Criteria:

1. Have had or simultaneously have other active malignant tumors within 5 years. Cured localized tumors, as basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, prostate carcinoma in situ, cervical carcinoma in situ, and breast in situ, are eligible;
2. Patients who are preparing for or have previously undergone organ or bone marrow transplantation;
3. Have ≥2 grade myocardial ischem or myocardial infarction, arrhythmia (QTc ≥470ms), and ≥2 grade congestive heart failure (New York Heart AssociationNYHA] classification);
4. Human immunodeficiency virus (HIV) infection;
5. Have active pulmonary tuberculosis;
6. Have a history or current presence interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, severe pulmonary dysfunction, etc., which may interfere with the detection and management of suspected drug-related pulmonary toxicity;
7. Have known active or suspected autoimmune diseases, except those in a stable state at the time of enrollment (not requiring systemic immunospressive therapy);
8. Have received live vaccine treatment within 28 days before the first dose; seasonal flu vaccines are not included;
9. Have received or need receive systemic corticosteroids (> 10 mg/day prednisone equivalent dose) or other immunosuppressive drugs within 14 days before the dose or during the study. However, the following cases are allowed: patients with no active autoimmune diseases can use topical or inhaled corticosteroids, or hormone replacement therapy with a dose ≤ 10 mg/day prednisone equivalent dose;
10. Have any active infection that requires systemic anti-infective within 14 days before the first dose; prophylactic antibiotic treatment (e.g., for urinary tract infections or chronic obstructive pulmonary disease) is not;
11. Have previously received other antibodies/drugs targeting immune checkpoints, such as PD-1, PD-L1, CTLA4, etc.;
12. Are currently receiving other clinical study treatments, or the time between the end of the previous clinical study treatment and the planned start of this study treatment is less than14 days;
13. Have a known severe allergic history to any monoclonal antibody or excipients of the study drug;
14. Have a history of psychiatric drug abuse or drug addiction; patients who have stopped drinking alcohol can be enrolled; According to the investigator's judgment, patients with serious concomitant that endanger the safety of the subjects or affect the completion of the study, or patients who are deemed unsuitable for enrollment for other reasons

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response rate (pCR) | 3 week

SECONDARY OUTCOMES:
The R0 resection rate after radical operation | 1 year
Major Pathological response (MPR) after radical operation | From baseline to after radical operation
Event Free Survival Rate from baseline to 1 year | from baseline to 1 year
Overall Survival rate from baseline to 1 year | From baseline to 1 year
Disease-related treatment failure rate from baseline to 1 year | From baseline to 1 year
Objective response rate from baseline to 1 year | From baseline to 1 year
Disease control rate from baseline to 1year | From baseline to 1year
Correlation between PD-L1 expression, TMB level and T cell subsets in tumour tissue samples and efficacy. | 6 week
The safety from baseline to 1year | From baseline to 1year

IPD SHARING:
Plan to Share IPD: No